CLINICAL TRIAL: NCT04759001
Title: Faecal Microbiota Transplantation to Eradicate Gut Colonisation From Carbapenem-resistant Enterobacteriaceae: a Randomised Controlled Trial
Brief Title: FMT for the Decolonization of Carbapenem-resistant Enterobacteriaceae
Acronym: FMT-CRE
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, IANIRO GIANLUCA, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3556
Record Dates: First submitted 2021-02-13; First posted 2021-02-17 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Enterobacteriaceae Infections; Multi-antibiotic Resistance
Keywords: Fecal microbiota transplantation; Enterobacteriaceae; Multi-drug resistant bacteria
MeSH Terms: conditions — Enterobacteriaceae Infections

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To mask treatments to physicisans and recipients, both FMT bottles and syringes will be covered with dark-coloured paper before the infusion, and the patients will be unable to see the endoscopic display during the procedure. Moreover, the physicians who will evsaluate patients at follow-up will not aware of the treatment being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Donor FMT (Experimental): Patients enrolled in this arm will receive donor FMT
  Interventions: Biological: Donor FMT
- Placebo FMT (Placebo Comparator): Patients enrolled in this arm will receive placebo FMT (that will be made of water)
  Interventions: Other: Placebo FMT

INTERVENTIONS:
Biological: Donor FMT — This intervention is represented by the administration, in the recipients' gut, of donor microbiota through FMT
  Arms: Donor FMT
Other: Placebo FMT — This intervention is represented by the administration, in the recipients' gut, of a placebo through FMT
  Arms: Placebo FMT

SUMMARY:
Rates of antimicrobial resistance are increasing worldwide. There is increasing evidence that physiological gut microbiota is a large reservoir of antibiotic-resistance genes. Healthy gut microbiota is known to prevent the colonization of the gastrointestinal tract by pathogens, the so-called mechanism of colonization resistance, but this protective mechanism can be altered by therapies that impair gut microbiota, including antibiotics or chemotherapeutics, with consequent colonisation of gut pathogens, including multi-drug resistant bacteria (MDRB). MDRB carriers represent an epidemiological threat to other hospitalized patients and to the whole community, but are also at risk of developing clinical consequences of this colonization, including bloodstream infections from these pathogens. Fecal microbiota transplantation (FMT) has shown high efficacy in the eradication of recurrent C. difficile infection, and initial evidence suggests that this procedure could be useful in eradicating also MDRB, mainly carbapenem-resistant Enterobacteriaceae.

However, current evidence is mostly limited to case reports and case series, and to a single randomised trial, which was stopped early and did not draw clear conclusion. In a systematic review of 21 studies and 192 patients, eradication rates ranged from 0% to 100%, and authors concluded that larger, well designed randomised controlled trials are needed to further explore this therapy.

The aim of this study is to investigate the efficacy of FMT, compared with placebo FMT, in eradicating gut colonisation from MDRB, focusing on CRE. The investigators will randomize patients colonized by CRE (diagnosed by rectal swab) to FMT from healthy donors or placebo, by colonoscopy. Then, patients will be followed up, rectal swabs will be repeated, and stool samples for culture and microbiome analysis will be collected, up to 3 months after FMT.

DETAILED DESCRIPTION:
Rates of antimicrobial resistance are increasing worldwide. There is increasing evidence that physiological gut microbiota is a large reservoir of antibiotic-resistance genes. Healthy gut microbiota is known to prevent the colonization of the gastrointestinal tract by pathogens, the so-called mechanism of colonization resistance, but this protective mechanism can be altered by therapies that impair gut microbiota, including antibiotics or chemotherapeutics, with consequent colonisation of gut pathogens, including multi-drug resistant bacteria (MDRB). MDRB carriers represent an epidemiological threat to other hospitalized patients and to the whole community, but are also at risk of developing clinical consequences of this colonization, including bloodstream infections from these pathogens. Fecal microbiota transplantation (FMT) has shown high efficacy in the eradication of recurrent C. difficile infection, and initial evidence suggests that this procedure could be useful in eradicating also MDRB, mainly carbapenem-resistant Enterobacteriaceae.

However, current evidence is mostly limited to case reports and case series, and to a single randomised trial, which was stopped early and did not draw clear conclusion. In a systematic review of 21 studies and 192 patients, eradication rates ranged from 0% to 100%, and authors concluded that larger, well designed randomised controlled trials are needed to further explore this therapy.

The extended aims of this study are:

* To compare the efficacy of donor FMT and placebo FMT in eradicating gut colonisation from CRE
* To compare the efficacy of donor FMT and placebo FMT in preventing clinical manifestations of gut colonisation from CRE
* To investigate changes in gut microbiome after treatments

The investigators will carry out a single-centre placebo-controlled, double blind randomised clinical trial of donor FMT vs placebo FMT in carriers of CRE Patients will be recruited among those referred to the infectious disease outpatient clinic of the Fondazione Policlinico Universitario "A. Gemelli". Patients with all inclusion criteria and none of the exclusion criteria (detailed in the specific section of this website) will be considered for this study.

Before randomisation, demographic data will be collected by the infectious disease staff. Moreover, patients will repeat rectal swab and stool culture.

Additionally, patients will be requested to give stool samples to be collected in a sterile, sealed container and stored at -80°C for metagenomic assessment of gut microbiome and meta-transcriptome assessment by the microbiology staff.

After baseline assessments, patients will be randomly assigned to one of the following treatment arms:

* Donor FMT (D-FMT)
* Placebo FMT (P-FMT)

Patients in both groups will undergo a single FMT procedure by colonoscopy. Each patient in the donor FMT group will receive faeces from one single donor. Placebo FMT will be made of 250 mL water. The selection of stool donors will be performed by the gastroenterology staff following protocols previously recommended by international guidelines and according the new recommendation imposed by the reorganisation of faecal microbiota transplant during the COVID-19 pandemic (Ianiro et al. - Gut 2020) The assignment of faecal infusates from healthy donors to patients will be done randomly, without any specific recipient-donor match, as this is not recommended by international guidelines All faecal infusates will be manufactured in the microbiology unit of our hospital. Only frozen faeces will be used. Preparation of frozen faeces will follow protocols from international guidelines.

Follow-up visits will be performed by physicians from the gastroenterology and the infectious disease unit. All patients will be followed up for 3 months after the end of treatments. Follow-up visits will be scheduled at week 1, week 2, week 4, and week 12, after the end of treatments, respectively. At each visit the following assessments will be performed: 1) rectal swab for MDRB; 2) collection of stool samples for stool culture ; 3) collection of stool samples for microbiome analysis; 4) record of adverse events. Unscheduled follow-up visits will be offered if requested by the patients.

Study Outcomes are detailed in the specific section of this website.

The statistical analysis will be performed both on an intention-to-treat and per-protocol basis. Differences among groups will be assessed with a two-tailed Wilcoxon-rank sum test for continuous data and with Fisher's exact probability test (using two-tailed P-values) for categorical data. Differences in cure percentages will be determined with Fisher's exact test (with two-tailed P values). For microbiome analysis, statistical differences between group means will be calculated using a two-tailed Wilcoxon-Rank Sum Test, through the R statistical software package (R Core Team, Vienna, Austria).

ELIGIBILITY:
Inclusion criteria

* 18 years old or older
* Current evidence of gut colonisation (diagnosed with rectal swab) by CRE
* Ability to give their consent to be included in the study.

Exclusion criteria

* Another known gastrointestinal infection apart from C. difficile infection
* Known active gastrointestinal disorders (e.g. infectious gastroenteritis, coeliac disease, inflammatory bowel disease, irritable bowel syndrome, chronic pancreatitis, biliary salt diarrhoea)
* Previous colorectal surgery or cutaneous stoma
* Food allergies
* Current or recent (<2 weeks) therapy with drugs that could possibly alter gut microbiota (e.g. antimicrobials, probiotics, proton pump inhibitors, immunosuppressants, metformin)
* Decompensated heart failure or heart disease with ejection fraction lower than 30%
* Severe respiratory insufficiency
* Psychiatric disorders
* Pregnancy
* Unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2025-02-18 (Actual); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Number of participants who will obtain an eradication of CRE carriage after treatments | 4 weeks
  The investigators will evaluate the number of participants who will obtain eradication of CRE carriage after treatments, at 4 weeks-follow-up, evaluated through rectal swab for CRE

SECONDARY OUTCOMES:
Number of participants who will obtain an eradication of CRE carriage after treatments | 12 weeks
  The investigators will evaluate the number of participants who will obtain eradication of CRE carriage after treatments, at 1,2 and 12 weeks-follow-up, evaluated through rectal swab for CRE
Number of participants with significant increase in alpha-diversity and beta-diversity of their gut microbiota after treatments | 12 weeks
  Throughout the study period (12 weeks) the investigators will evaluate the number of participants with significant increase in alpha-diversity (assessed by Shannon index) and beta-diversity (assessed by Bray-Curtis dissimilarity) of their gut microbiota after treatments, compared with baseline
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 12 weeks
  The number of participants with treatment-related adverse events (assessed by CTCAE v4.0) will be recorded throughout the study period (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Ianiro, Principal Investigator — Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Digestive Disease Center, Fondazione Policlinico Univesitario A. Gemelli IRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available to other researchers
Supporting Information: Study Protocol
Time Frame: data will be available after the completion of the study, for 5 years
Access Criteria: Data will be given upon reasonable request to the PI

REFERENCES:
- [Background] Pitout JD, Laupland KB. Extended-spectrum beta-lactamase-producing Enterobacteriaceae: an emerging public-health concern. Lancet Infect Dis. 2008 Mar;8(3):159-66. doi: 10.1016/S1473-3099(08)70041-0. PMID 18291338
- [Background] Huttner BD, de Lastours V, Wassenberg M, Maharshak N, Mauris A, Galperine T, Zanichelli V, Kapel N, Bellanger A, Olearo F, Duval X, Armand-Lefevre L, Carmeli Y, Bonten M, Fantin B, Harbarth S; R-Gnosis WP3 study group. A 5-day course of oral antibiotics followed by faecal transplantation to eradicate carriage of multidrug-resistant Enterobacteriaceae: a randomized clinical trial. Clin Microbiol Infect. 2019 Jul;25(7):830-838. doi: 10.1016/j.cmi.2018.12.009. Epub 2019 Jan 4. PMID 30616014
- [Background] Cammarota G, Ianiro G, Kelly CR, Mullish BH, Allegretti JR, Kassam Z, Putignani L, Fischer M, Keller JJ, Costello SP, Sokol H, Kump P, Satokari R, Kahn SA, Kao D, Arkkila P, Kuijper EJ, Vehreschild MJG, Pintus C, Lopetuso L, Masucci L, Scaldaferri F, Terveer EM, Nieuwdorp M, Lopez-Sanroman A, Kupcinskas J, Hart A, Tilg H, Gasbarrini A. International consensus conference on stool banking for faecal microbiota transplantation in clinical practice. Gut. 2019 Dec;68(12):2111-2121. doi: 10.1136/gutjnl-2019-319548. Epub 2019 Sep 28. PMID 31563878
- [Background] Ianiro G, Mullish BH, Kelly CR, Kassam Z, Kuijper EJ, Ng SC, Iqbal TH, Allegretti JR, Bibbo S, Sokol H, Zhang F, Fischer M, Costello SP, Keller JJ, Masucci L, van Prehn J, Quaranta G, Quraishi MN, Segal J, Kao D, Satokari R, Sanguinetti M, Tilg H, Gasbarrini A, Cammarota G. Reorganisation of faecal microbiota transplant services during the COVID-19 pandemic. Gut. 2020 Sep;69(9):1555-1563. doi: 10.1136/gutjnl-2020-321829. Epub 2020 Jul 3. PMID 32620549
- [Background] Saha S, Tariq R, Tosh PK, Pardi DS, Khanna S. Faecal microbiota transplantation for eradicating carriage of multidrug-resistant organisms: a systematic review. Clin Microbiol Infect. 2019 Aug;25(8):958-963. doi: 10.1016/j.cmi.2019.04.006. Epub 2019 Apr 12. PMID 30986562